CLINICAL TRIAL: NCT00805636
Title: Evaluation of Efficacy and Safety of 18FML10, as a PET Imaging Radiotracer, in Early Detection of Response of Brain Metastases of Non-Hematological Solid Tumors to Radiation Therapy
Brief Title: Evaluation of the Efficacy and Safety of [18F]-ML-10, as a PET Imaging Radiotracer, in Early Detection of Response of Brain Metastases of Solid Tumors to Radiation Therapy.
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Aposense Ltd. (Industry)
Responsible Party: Miri Ben-Ami, MD, Aposense
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: NST-CA004CTIL
Record Dates: First submitted 2008-12-07; First posted 2008-12-09 (Estimated); Last update posted 2010-05-12 (Estimated); Status verified 2010-04

CONDITIONS: Brain Metastases; Solid Tumors
Keywords: cell death; PET imaging; brain metastases; stereotactic radiosurgery
MeSH Terms: conditions — Brain Neoplasms | interventions — 5-fluoropentyl-2-methylmalonic acid; Spermine Synthase; Therapeutics; Magnetic Resonance Spectroscopy

INTERVENTIONS:
Drug: 2-(5-fluoro-pentyl)-2-methyl-malonic-acid ([18F]-ML-10) — [18F]-ML-10 will be radiolabeled at the PET Radioactive Drug Production (RDP) facility at or in close proximity to each clinical site, and will be administered as an intravenous bolus injection (in 3-10 ml sterile saline solution, containing no more than 10% ethanol by volume). The dose concentration selected for [18F]-ML-10 will be 7 MBq/Kg or 0.19 mCi/Kg. The radioactivity dosage of [18F]-ML-10 administered at each PET/CT session will be at least 300 MBq (8.1 mCi) and not more than 500 MBq (13.5 mCi).
  Other Names: [18F]-ML-10
Radiation: Stereotactic Radio-Surgery (SRS) therapy — SRS will be administered according to the standard of care using a radiation dose of 14-24 Gy to each lesion.
Procedure: Positron Emission Tomography — Each patient will undergo 2 PET/CT sessions, each following intravenous administration of [18F]-ML-10, to assess tracer uptake by the brain metastases treated by SRS. The PET/CT scan will be directed to the brain and will include one bed position. The PET/CT sessions will be performed at baseline, i.e., before the radiation treatment, and on the day after, within 24h after SRS treatment.

SUMMARY:
The purpose of this study is to evaluate the potential of [18F]-ML-10 to serve as an imaging tool for the early detection of response of brain metastases to radiation therapy. Such early detection may help early identification of responsive and non-responsive lesions. The experimental design of the present study aims to evaluate the potential of PET imaging with [18F]-ML-10 to address the currently unmet clinical need for very early (within one day)assessment of response to therapy. Currently, response assessment is available only after several weeks or months after completion of therapy, when tumor shrinkage can be detected by anatomical imaging (by MRI). Early detection of tumor response to treatment is now widely-recognized as a highly-desirable goal in oncology, and is respectively the target of intense research worldwide. In the future, the option to know early upon treatment administration, that the treated tumor is a non-responsive, may improve clinical management of patients with brain metastases of solid tumors.

DETAILED DESCRIPTION:
Early assessment of the efficacy of anti-cancer therapy is highly desirable and an unmet need in clinical oncology. Currently, treatment efficacy is mostly measured by following tumor size by anatomical imaging (CT scan or MRI). However, changes in tumor size may be observed only after several weeks to several months after completion of treatment. Meanwhile, in cases where there is no response, the patient is unnecessarily exposed to treatment's side effects, and precious time may be lost before the initiation of an alternative, potentially more beneficial line of therapy. Therefore, there is an urgent and serious need for better tools for monitoring of tumor response to anti-cancer treatments.

To address this need, [18F]-ML-10, a novel small molecular-weight probe (MW 205) was developed for clinical detection of apoptosis in vivo by positron emission tomography (PET). [18F]-ML-10 is a member of the Aposense family of compounds, a novel class of molecular probes for molecular imaging of cell death. The proposed indication for which [18F]-ML-10 is being developed is for early assessment of response of solid tumors to radiation and chemoradiation therapy.

Previous preclinical and clinical studies have substantiated the safety of [18F]-ML-10, its very high stability in vivo, its favorable biodistribution profile, and its efficacy in clinical detection of cell death. In preclinical studies, the selective retention of [18F]-ML-10 in the focus of the neurovascular cell death in cerebral ischemia was demonstrated in respective animal models. [18F]-ML-10 has been examined in two clinical trials in Uppsala Imanet, Sweden, and has been found safe in administration to healthy subjects and to elderly subjects with acute ischemic cerebral stroke. In these clinical trials, [18F]-ML-10 was also found efficacious in the clinical imaging of apoptosis, being either physiological apoptosis as observed in the testes in young healthy males, and pathological cell death, as observed in the brains of patients with acute ischemic cerebral stroke.

Additional Phase 2 study demonstrated the suitability and safety of 18F-ML-10, designed to serve as a PET radiotracer for early detection of cellular apoptosis of brain metastases in response to WBRT. The relationship between the early change in 18F-ML-10 uptake by the tumor, observed during or upon completion of treatment, and subsequent tumor shrinkage as observed by MRI eight weeks after the completion of WBRT, was demonstrated.18F-ML-10 demonstrated a good safety profile with no drug-related AEs or any effect on safety parameters.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female patients with metastatic non- hematological solid tumors, with one or more brain metastases, of which at least one lesion has a diameter ≥1.5 cm, as confirmed by anatomical imaging (GBCA-enhanced MRI), wherein this lesion (or lesions) is scheduled to be treated by SRS.
2. ECOG performance status of 0, 1 or 2 at the time of enrollment.
3. Women of child-bearing potential must have a negative blood pregnancy test at screening and use an adequate and medically acceptable contraceptive method.
4. Willing and able to follow the protocol requirements.
5. Able to provide written informed consent.

Exclusion Criteria:

1. Unstable medical condition, such as ischemic heart disease, or any other disease or medical condition that may place the patient at added risk during the study, as assessed by the Principal Investigator. A patient with a seizure disorder, focal or generalized, not adequately controlled by anti-convulsant therapy, and /or patient who have experienced an event of focal or generalized seizure within 7 days prior to screening will be considered neurologically unstable.
2. Any indication of a risk for an imminent brain herniation, as evaluated by the Principal Investigator, based on the findings on brain MRI.
3. Treatment with whole brain radiation therapy (WBRT) within 3 months prior to screening.
4. Evidence for hemorrhage within any of the brain metastases.
5. Any known psychiatric disorder other than mild depression or anxiety that may affect adherence to the study requirements.
6. Known allergy to gadolinium.
7. Any contraindication to MR imaging (e.g., metal implant, aneurysm clip, pacemaker).
8. Other condition that, in the opinion of the Investigator, might jeopardize the safety of the patient, or the adequate evaluation of study results.
9. Treatment with any investigational drug, device or biologic agent within 30 days prior to administration of [18F]-ML-10.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2008-11; Primary Completion 2010-10 (Estimated); Study Completion 2010-10 (Estimated)

PRIMARY OUTCOMES:
To assess the relationship between changes in 18FML10 uptake in the target lesions (PET/CT) obtained before and after radiotherapy (SRS), and changes of the lesions size (MRI, ~8w after SRS) in response to treatment, according to the WHO criteria | 1 year

SECONDARY OUTCOMES:
Characterization of early alterations in the voxel-based 18FML10 uptake in the target lesion in response to the single fraction high-dose Stereotactic RadioSurgery, SRS. 18FML10 uptake at 24h after SRS and at baseline, before SRS, will be compared | 1 year
To identify parameters derived from the changes in 18FML10 uptake observed early after SRS that can discriminate responsive from non-responsive target lesions, and to estimate optimal cut-off values of this parameter (sensitivity and specificity) | 1 year
To perform additional analyses for all other lesions with longest diameter ≥ 1.5 cm treated by SRS. | 1 year

CONTACTS AND LOCATIONS:
Locations (4):
- United States (4):
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - Department of Radiation oncology, Memorial Sloan Kettering Cancer Center, New York, New York
  - UPMC Shadyside Radiation Oncology, Pittsburgh, Pennsylvania